CLINICAL TRIAL: NCT05361993
Title: Efficacy of Biofeedback in the Treatment of Tic Disorder：A Randomized Controlled Trial
Brief Title: Efficacy of Biofeedback in the Treatment of Tic Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been temporarily halted due to a malfunction with the biofeedback equipment we are using. At present, we do not have the necessary funds to repair the equipment, and as a result, the research has been suspended for the time being.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Normal University (Unknown)
Responsible Party: Principal Investigator, Ding Qiang, Clinical Psychotherapist, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TD_BF_RCT20220318
Record Dates: First submitted 2022-03-18; First posted 2022-05-05 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Tic Disorders
Keywords: biofeedback; drug therapy; Clinical Efficacy; Cognitive flexibility
MeSH Terms: conditions — Tic Disorders | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofeedback therapy (Experimental): three times a week, every other day interval, 30 minutes each time, each subject received 20 biofeedback training (using the Infiniti3000A biofeedback system Patients in the theta group decreased the theta amplitude at Cz. Patients in the theta group received positive feedback when their theta activity was below the feedback threshold.
  Interventions: Device: biofeedback
- Drug therapy (Active Comparator): Considering the patients with chronic tic disorder (chronic motor or vocal tic disorder or Tourette's disorder), aripiprazole was selected as a single drug with constant dose during the treatment. In case of extrapyramidal side effects, benhexol was given to reduce the extrapyramidal side effects, and the dosage and duration of medication were recorded
  Interventions: Drug: Drug Aripiprazole

INTERVENTIONS:
Drug: Drug Aripiprazole — Considering the patients with chronic tic disorder (chronic motor or vocal tic disorder or Tourette's disorder), aripiprazole was selected as a single drug with constant dose during the treatment. In case of extrapyramidal side effects, benhexol was given to reduce the extrapyramidal side effects, and the dosage and duration of medication were recorded
  Arms: Drug therapy
Device: biofeedback — Biofeedback therapy Biofeedback therapy, three times a week, every other day interval, 30 minutes each time, each subject received 20 biofeedback training（using the Infiniti3000A biofeedback system，Thought Technology Ltd.）.Patients in the theta group decreased the theta amplitude at Cz. Patients in the theta group received positive feedback when their theta activity was below the feedback threshold.
  Arms: Biofeedback therapy

SUMMARY:
To investigate the efficacy of EEG biofeedback and drug therapy in the treatment of tic disorders

DETAILED DESCRIPTION:
This study intends to investigate the efficacy of EEG biofeedback and drug therapy on clinical symptoms, cognitive flexibility and quality of life in chronic tic disorder and Tourette syndrome through a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders(Fifth Edition,DSM-5) for chronic tic disorder or Tourette syndrome（TS）;
* Ethnic group is Han nationality;
* Aged 8 ~ 16 years old;
* otal IQ of Wechsler Intelligence Scale for Children ≥ 80 points for subjects;
* Symptom severity score in Yale Global Severity Scale (YGTSS), TS patients > 13, CTD > 9;
* Did not receive any drug (including traditional Chinese medicine) treatment 4 weeks before enrollment;
* Obtain written informed consent from children and guardians

Exclusion Criteria:

* Epilepsy, cardiovascular disease
* Patients with schizophrenia, mental retardation, autism spectrum disorder, bipolar disorder and major depression who meet the DSM-5 diagnostic criteria;
* Receiving systematic traditional Chinese medicine treatment one month before enrollment or currently;
* Receiving systematic psychotherapy one month before enrollment or currently;
* Receive systematic physical therapy one month before enrollment or currently
* Those who cannot follow the doctor's advice or refuse to cooperate;
* Those with obvious abnormal laboratory test results (AST or ALT ≥ 2 times of the upper limit of normal value; bun ≥ 1.5 times of the upper limit of normal value; Cr ≥ 1.2 times of the upper limit of normal value);
* Prolongation of QTc interval (QTc ≥ 450 ms in men or ≥ 470 MS in women);

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Yale global tic severity scale | baseline assessment (T0)
  Tic symptom severity is estimated by Yale Global Tic Severity Scale Total Tic score. The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics-scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.Lower scores indicate improvement and higher scores indicate worsening.
Yale global tic severity scale | assessment after 4 weeks of treatment (T1)
  Tic symptom severity is estimated by Yale Global Tic Severity Scale Total Tic score. The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics-scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.Lower scores indicate improvement and higher scores indicate worsening.
Yale global tic severity scale | assessment after 8 weeks of treatment (T2)
  Tic symptom severity is estimated by Yale Global Tic Severity Scale Total Tic score. The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics-scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.Lower scores indicate improvement and higher scores indicate worsening.
Yale global tic severity scale | 3-month follow-up after completion of treatment (T3).
  Tic symptom severity is estimated by Yale Global Tic Severity Scale Total Tic score. The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics-scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.Lower scores indicate improvement and higher scores indicate worsening.
Wisconsin Card Sorting Test | baseline assessment (T0)
  The participants were asked to sort 64 cards to match either color (red, blue, yellow, or green), form (crosses, circles, triangles, or stars), or number of figures (one, two, three, four). During the task, the sorting rule changed discreetly from color to form or number of figures without the participants being informed. The participants had to shift sets accordingly and sort cards following the new sorting rule. Set shifting difficulties were indicated by preservative errors; thus, higher scores on this test represent worse performance.
Wisconsin Card Sorting Test | assessment after 4 weeks of treatment (T1)
  The participants were asked to sort 64 cards to match either color (red, blue, yellow, or green), form (crosses, circles, triangles, or stars), or number of figures (one, two, three, four). During the task, the sorting rule changed discreetly from color to form or number of figures without the participants being informed. The participants had to shift sets accordingly and sort cards following the new sorting rule. Set shifting difficulties were indicated by preservative errors; thus, higher scores on this test represent worse performance.
Wisconsin Card Sorting Test | assessment after 8 weeks of treatment (T2)
  The participants were asked to sort 64 cards to match either color (red, blue, yellow, or green), form (crosses, circles, triangles, or stars), or number of figures (one, two, three, four). During the task, the sorting rule changed discreetly from color to form or number of figures without the participants being informed. The participants had to shift sets accordingly and sort cards following the new sorting rule. Set shifting difficulties were indicated by preservative errors; thus, higher scores on this test represent worse performance.
Wisconsin Card Sorting Test | 3-month follow-up after completion of treatment (T3)
  The participants were asked to sort 64 cards to match either color (red, blue, yellow, or green), form (crosses, circles, triangles, or stars), or number of figures (one, two, three, four). During the task, the sorting rule changed discreetly from color to form or number of figures without the participants being informed. The participants had to shift sets accordingly and sort cards following the new sorting rule. Set shifting difficulties were indicated by preservative errors; thus, higher scores on this test represent worse performance.

SECONDARY OUTCOMES:
Color-word Stroop task | It's a repeated measurement variable，baseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  The Stroop task requires participants to name the ink color of a series of color words. In the congruent condition, the color name corresponds exactly to the color of each letter; in the incongruent condition, the printed word and the actual color of each letters are different. When subjects are required to report the ink color of the word, greater difficulty is experienced when they are in the incongruent condition. This difficulty can be measured by the increase in the amount of time required to complete the task (the Stroop interference effect). The measure of executive ability is the relative response delay in the Stroop interference condition as measured by response time (RT) in the incongruent condition minus RT in the neutral condition.
The Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) | It's a repeated measurement variable，baseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  The CY-BOCS evaluates the severity of obsessions and compulsions, using ten items across five dimensions (time occupied by symptoms, interference, distress, resistance and degree of control over symptoms). The total severity score can range from 0 to 40. CY-BOCS total scores in the range of 14-24 are considered moderate, 25-30 moderate-severe and over 30 severe
The parent version of Swanson, Nolan, and Pelham-IV(SNAP-IV) | It's a repeated measurement variable，baseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  It contains 26 items and is scored on a 0-3 Likert scale. The scale consists of three subscales, which are three parts: attention deficit, hyperactivity/impulsivity, and oppositional defiance, and can be used for the assessment of ADHD symptoms in tic symptom comorbidity in this study.
Children' s Depression Inventory(CDI) | It's a repeated measurement variable，baseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  There are 27 items quantifying symptoms such as depressed mood, hedonic capacity, vegetative functions, self-evaluation, and interpersonal behaviors. Each item consists of three statements graded in order of increasing severity from 0 to 2; children and adolescents select the one that characterized their symptoms best during the past 2 weeks. The item scores are combined into a total depression score, which ranges from 0 to 54. A higher CDI score means a higher depressive state.
The Screen for Child Anxiety Related Emotional Disorders(SCARED) | It's a repeated measurement variable，aseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  The SCARED is a 41-item self-report measure designed to screen for DSM-IV anxiety disorders. The SCARED includes 5 factors: somatic/panic (13 items; e.g., "When I feel frightened, it is hard to breathe"), generalized anxiety (9 items; e.g., "I worry about other people liking me"), separation anxiety (8 items; e.g., "I get scared if I sleep away from home"), social phobia (7 items; e.g., "I don't like to be with people I don"t know well"), and school phobia (4 items; e.g., "I get headaches when I am at school"). The participants rated the items of each factor on a 3-point scale (0 = not true or hardly ever true, 1 = sometimes true, and 2 = true or often true). The SCARED total score, derived by adding the responses of the 41 items, ranges from 0 to 82.
Conners' Parent Rating Scale-Revised（CPRS-R） | It's a repeated measurement variable，aseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  It is suitable for children aged 3 - 16 years, and a total of 48 items in this scale include six factors: conduct problems, learning problems, psychosomatic problems, impulsive-hyperactivity, anxiety, and hyperactivity index, with a total of 48 items, which are scored on a 0-3 four-level scale.
The Clinical Global Impression-severity scale | It's a repeated measurement variable，baseline assessment (T0), assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  The severity of illness subscale is designed to acquaint the patient's severity of symptoms with those of other people experiencing the same mental ailment. The CGI-S rates this severity of a 1-7 scale, with (1) representing normal symptoms, meaning the patient is not ill. The highest on the scale, (7), represents patients among the most severely ill. Right in the middle at (4), a patient will be defined as moderately ill.
Clinical Global Impressions-Improvement scale | It's a repeated measurement variable，assessment after 4 weeks of treatment (T1), assessment after 8 weeks of treatment (T2), and 3-month follow-up after completion of treatment (T3)
  The global improvement subscale allows the practitioner to create a comparative improvement based on the baseline of the first test. These changes reflect how symptoms have or have no improves due to treatment. The 7-point CGI-I scale rates improvement with a (1) representing a 'very much improved' patient and (7) representing a patient who has become 'very much worse' due to treatment. The rating (4) represents a patient displaying no change from the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fundan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No